CLINICAL TRIAL: NCT04614285
Title: Partial Excavation of Dentin Carious Lesions in Primary Molars: A Practice-Based Research Network (PBRN) Study
Brief Title: Partial or Complete Excavation of Deep Caries in Primary Molars
Acronym: PBRN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Annika Julihn, DDS, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnr. 2018/743-31/1
Record Dates: First submitted 2020-06-15; First posted 2020-11-03 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Dental Caries in Children
Keywords: Dental caries; Dental treatment; Pediatric dentistry; Practice-based research network; Randomized clinical trial
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: The study has a prospective multi-center, two arms randomized controlled clinical trial design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial excavation (Experimental): The treatment will be performed after applying local anesthetic according to individual needs. The intervention group will receive partial removal of the carious lesion; In the inner part of the lesion, the caries removal will be limited to reach leathery or slightly soft dentin by probing. The restorations will be placed according to evidence based methods and the material used according to the operators material of choice.
  Interventions: Procedure: Partial excavation
- Complete excavation (Active Comparator): The treatment will be performed after applying local anesthetic according to individual needs. The control group will receive the same treatment procedure as the intervention group, but the excavation procedure will include total removal of the carious tissue. The total caries removal will be ensured with hardness on probing and the visual examination. Photographs will be used as benchmark.
  Interventions: Procedure: Partial excavation

INTERVENTIONS:
Procedure: Partial excavation — Operators sign up for participation at the homepage of Center for Pediatric Oral Health Research (ABC). The study will be carried out in a Practice-Based Research Network setting. All practitioners interested in participating in the study will get access to an online information about their participation after they signed up. The participation starts by answering a questionnaire on their treatment attitudes and experiences.
  Patients will be identified during the routine dental examination. If a carious lesion in the primary molars is detected and in a need of a restoration, the children and parents will be asked to participate in the study.
  The parents receive information about the study and give their consent. Allocation into treatment groups will be performed by random assignment by the homepage of ABC.
  After the study is finished the participating dentist will be asked to answer the same questionnaire to investigate the effect of the participation on the operators attitude.
  Other Names: Selective excavation; Incomplete excavation

SUMMARY:
Background: The traditional approach of carious lesions with risk for progression has has been to excavate all infected and demineralised tissue before placement of the restoration. In primary teeth, treatment of deep carious lesions is associated with significant risk of pulp lesions and postoperative complications and thus the risk of the teeth being lost. During the past decade, more focus has been on biological methods for caries excavating of deep dentin lesions. An overview comparing different biological methods such as partial or stepwise excavation of deep dentin caries in primary teeth shows that they work as well as traditional methods performing complete caries excavation but have the benefits of reducing the risk of iatrogenic pulp damage [1-3].

Our primary hypothesis is that there is no difference in tooth or filling survival after partial caries excavation compared to complete caries excavation in primary molars.

The secondary hypothesis is that the therapist's knowledge, experience and treatment attitudes and choices are not affected by a participation in the study.

DETAILED DESCRIPTION:
The treatment of carious lesions with risk for progression has traditionally been done with caries removal and restorative treatment of the affected teeth. In primary teeth, different treatments for deep carious lesions have been described. Complete excavation aims to removing all infected and demineralised dentin with a high risk of pulpal exposure, postoperative complications and thus the risk of the teeth being lost. In many cases, treatment also involves pain and suffering for the patient, which can lead to dental fear among children.

In latest years there has been a growing evidence for the possibility of controlling the cariogenic biofilm in the lesion by isolating the infected tissue from the oral cavity with an isolating restoration and leaving infected tissue under the permanent restoration. The methods are considered to be able to slow down or arrest the caries progression in primary teeth so that the teeth exfoliate without causing pain or infection. When carious tissue is isolated from the oral environment deprives the residual bacteria from carbohydrates and has thus been shown to have an antibacterial effect and to stop further progression of the lesion [4-5]. Partial, i.e. one-step incomplete or selective excavation is one biological method that seals carious dentin under a definitive restoration, omitting any re-entry. This can thus be a treatment choice for the primary teeth.

An overview comparing different biological methods for caries excavation of deep dentin caries in primary teeth, such as partial or stepwise excavation shows that they work as well as traditional methods performing complete caries excavation but have the benefits of reducing the risk of iatrogenic pulp damage [1-4]. However, partial excavation compared with complete excavation in deep carious lesions in primary teeth has not previously been tested under practice-like conditions. If the study shows that the treatment is effective in clinical practice and in the hands of multiple operators, it will change the routine treatment of dentin caries in primary teeth, thus increasing the survival of teeth and fillings, as well as reducing the risk of unwanted injury to the pulp and pain and discomfort to the children.

Objectives and Hypothesis: The primary purpose of the study is to investigate the sustainability of filling and the tooth survival after two different methods of excavation of dentin caries in primary molars.

The primary hypothesis is that there is no difference in tooth or filling survival after partial caries excavation compared to complete caries excavation in primary molars.

The secondary purpose of the study is to investigate the therapist's knowledge, experience and treatment attitude and choice of treatment method in primary caries excavation and how a participation in the study affects the therapist.

The secondary hypothesis is that the therapist's knowledge, experience and treatment attitudes and choices are not affected by a participation in the study.

The study aims to testing a newly started Practice-Based Research Network (PBRN) within the discipline of pediatric dentistry in the Stockholm city county in Sweden and the county of Östergötland. Thus, the scientific question will be tested under an effectiveness setting including practitioners interested in participating in the PBRN by signing up for participating in this particular study. The study has a prospective multi-center, two arms randomized controlled clinical trial design.

ELIGIBILITY:
Inclusion Criteria:

* Children in the age of 3-8 years, with one or more primary molar teeth in a need of a restoration due to a moderate depth of carious lesion;

  * caries lesion diagnosed into dentin on radiographs though not exceeding the inner third of the dentin
  * caries lesion diagnosed visually with a cavity into dentin.

Exclusion Criteria:

* Children with behaviour management problems.
* Teeth with pulpal symptoms
* Teeth expected to exfoliate within the next 18 months

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Success | 24 months
  Success will be measured by assessing if the restoration is in place (i.e. tooth in place vs. tooth lost) and without comment.
Tooth survival | 24 months
  Tooth survival will be measured by assessing tooth exfoliation without causing pain or infection.

SECONDARY OUTCOMES:
Decision-making Questionnaire | 24 months
  The Dentist's Knowledge and Attitudes of Deep Carious Lesions in Primary Teeth questionnaire will be used to assess dentists' knowledge, experience, treatment and attitudes and how these factors were affected by participation in the study. The questionnaire is rated on a scale from 1-4, with 1 having the least impact or what the dentist does most rarely, and 4 having the the greatest impact or what the dentist does most often. The questionnaire will be administered at baseline and at 24-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Göran Dahllöf, Professor, Principal Investigator — Department of Dental Medicine, Karolinska Institutet, Sweden
Locations (1):
- Division of Orthodontics and Pediatric Dentistry, Department of Dental Medicine, Karolinska Institutet, Sweden, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franzon R, Guimaraes LF, Magalhaes CE, Haas AN, Araujo FB. Outcomes of one-step incomplete and complete excavation in primary teeth: a 24-month randomized controlled trial. Caries Res. 2014;48(5):376-83. doi: 10.1159/000357628. Epub 2014 Apr 8. PMID 24732081
- [Background] Griffin SO, Oong E, Kohn W, Vidakovic B, Gooch BF; CDC Dental Sealant Systematic Review Work Group; Bader J, Clarkson J, Fontana MR, Meyer DM, Rozier RG, Weintraub JA, Zero DT. The effectiveness of sealants in managing caries lesions. J Dent Res. 2008 Feb;87(2):169-74. doi: 10.1177/154405910808700211. PMID 18218845
- [Background] Oong EM, Griffin SO, Kohn WG, Gooch BF, Caufield PW. The effect of dental sealants on bacteria levels in caries lesions: a review of the evidence. J Am Dent Assoc. 2008 Mar;139(3):271-8; quiz 357-8. doi: 10.14219/jada.archive.2008.0156. PMID 18310731
- [Result] Ricketts D, Lamont T, Innes NP, Kidd E, Clarkson JE. Operative caries management in adults and children. Cochrane Database Syst Rev. 2013 Mar 28;(3):CD003808. doi: 10.1002/14651858.CD003808.pub3. PMID 23543523
- [Result] Schwendicke F, Dorfer CE, Paris S. Incomplete caries removal: a systematic review and meta-analysis. J Dent Res. 2013 Apr;92(4):306-14. doi: 10.1177/0022034513477425. Epub 2013 Feb 8. PMID 23396521